CLINICAL TRIAL: NCT01876771
Title: An Open-label Phase II Study of Lutetium-177 [DOTA0, Tyr3] Octreotate (Lu-DOTA-TATE) Treatment in Patients With Somatostatin Receptor Positive Tumours
Brief Title: A Trial to Assess the Safety and Effectiveness of Lutetium-177 Octreotate Therapy in Neuroendocrine Tumours
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TX-LUT-001; HREBA.CC-18-0165 (Other: Health Research Ethics Board of Alberta Cancer Committee)
Record Dates: First submitted 2013-04-10; First posted 2013-06-13 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Carcinoma, Neuroendocrine
Keywords: 177lutetium-DOTA(O)Tyr3)octreotate
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [177]Lu-DOTA-TATE Therapy (Experimental): Nominal, induction stage dose of 150 mCi (5.55 GBq) [177]Lu-DOTA-TATE every 10 - 14 weeks for 4 treatments.
  Nominal maintenance stage dose of 100 mCi (3.7 GBq) [177]Lu-DOTA-TATE every 22 - 40 weeks, up to a maximum of 8 treatments.
  Interventions: Drug: [177]Lu-DOTA-TATE

INTERVENTIONS:
Drug: [177]Lu-DOTA-TATE — Peptide receptor radionuclide therapy (PPRT)
  Other Names: Lu-DOTA-TATE

SUMMARY:
Neuroendocrine tumours (NETs) are rare, slow growing, and diagnosis is often delayed with advanced metastases at presentation. In select patient populations, radioisotope therapy with Lutetium-177 (Lu-DOTA-TATE) has been shown to be a safe and effective palliative therapy, and has been widely used by research groups in Europe. A brand of Lu-DOTA-TATE (Lutathera(R)) is approved for the treatment of gastroenteropancreatic NETs in Europe, the U.S., and more recently in Canada. While Lutathera(R) is approved in Canada, it is not publicly funded in Alberta. Lu-DOTA-TATE has been used at the Cross Cancer Institute to treat more than 300 patients with NETs since August, 2010. Our Lu-DOTA-TATE treatment was initially given under Health Canada's Special Access Programme (SAP), with each individual treatment requiring separate approval. In 2014, Health Canada requested we conduct a clinical trial with Lu-DOTA-TATE instead.

The purpose of this study is to: 1) assess the efficacy of Lu-DOTA-TATE treatment in patients with somatostatin receptor positive tumours; 2) assess the safety of Lu-DOTA-TATE; 3) assess the effect of Lu-DOTA-TATE on Quality of Life and survival.

DETAILED DESCRIPTION:
The proposed clinical trial will be a Phase II, open label, single site study in subjects with somatostatin receptor positive tumours. Radioactive Lu-DOTA-TATE doses are fixed within a range of 1.85 - 5.55 GBq ± 10%, with individual doses based on specified risk factors. There will be two groups of subjects enrolled in this study. Group A subjects (primary therapy) will have progressive somatostatin receptor positive tumours and have never received Lu-DOTA-TATE. Group B subjects (maintenance therapy) will be those subjects who have previously received Lu-DOTA-TATE under the Special Access Programme (SAP) and will maintain their treatment schedule when they are entered into the study.

All subjects in Group A will be treated in an induction stage using 10-14 week dosing for up to 4 treatments. If an individual patient shows stable or improving disease status with no significant toxicities after the 4 induction treatments, they will be assessed 12-20 weeks after the last therapeutic treatment for entry into the maintenance stage. Patients will be re-assessed for stable or improving disease status with no significant toxicities 12-20 weeks after every other treatment of the maintenance stage for consideration of further maintenance treatments (re-evaluations), up to a maximum of 8 treatments per patient if there have been no significant toxicities or progression. At each treatment, an amino acid solution is infused prior to and during the Lu-DOTA-TATE infusion to protect the kidneys. Subjects will be followed for 6 months and 1 year (± 4 weeks) following their last treatment dose to determine progression-free survival, and annually (± 4 weeks) for up to 5 years following their last treatment dose to determine overall survival. All subjects meeting evaluation criteria will be analysed for safety, and all Group A subjects who have received at least two treatments of Lu-DOTA-TATE will be evaluated for efficacy. Those Group B subjects with adequate baseline data for comparison collected retrospectively from a chart review study (REV-LUT-001) may also be evaluated for safety and efficacy. Additional optional characterization of tumour samples from subjects who have had surgery before or during the study may be performed to characterize NET tumour biology changes following Lu-DOTA-TATE treatment.

ELIGIBILITY:
Group A (Primary Therapy) Inclusion Criteria:

1. Male or female ≥ 14 - 90 years of age.
2. At least 1 tumour site reliably evaluable by CT or magnetic resonance imaging (MRI) of at least 1.0 cm (smallest dimension) or ≥ 1.5 cm lymph node disease (smallest dimension) (the target lesion) within 26 weeks of enrolment, with documented presence of somatostatin receptors on radionuclide imaging, with uptake greater than liver background as assessed by planar Octreoscan® images or Ga-68 labelled somatostatin analogue (68Ga-DOTATATE or 68Ga-HA-DOTATATE) PET imaging (or other available somatostatin receptor targeting PET agents) obtained within 1 year of enrolment. Patients with bone-only disease can be enrolled provided there is presence of somatostatin receptor positive tumour(s) on radionuclide imaging corresponding to osteolytic or osteoblastic bone lesions on CT or MRI, with uptake greater than liver background as assessed by planar Ocgtreoscan(R) images or somatostatin receptor PET imaging regardless of size.
3. Histologically confirmed diagnosis of neuroendocrine tumor.
4. Progressive disease documented by anatomic imaging and/or presence of new lesions on somatostatin receptor imaging assessed by comparable studies. In the opinion of the investigator, patients with no progression on imaging may still be considered eligible in presence of carcinoid symptoms refractory to treatment with somatostatin receptor analogues or functional Pheochromocytoma/Paraganglioma symptoms that are not well controlled with current medical treatment.
5. 18F-FDG PET/CT whole-body imaging within 26 weeks of enrolment.
6. Life expectancy greater than 12 weeks from enrollment.
7. Serum creatinine ≤ 150 µmol/L, and a calculated (Cockcroft-Gault) or estimated GFR of ≥ 50 mL/min measured within 2 weeks of enrollment.
8. Haemoglobin concentration ≥ 90 g/L; white blood cell (WBC) count ≥ 2 x 10^9/L; platelets ≥ 100 x 10^9/L measured within 2 weeks of enrolment.
9. Liver function tests (total bilirubin, alanine transaminase (ALT), aspartate transaminase (AST)) ≤ 3X the limit of normal measured within 2 weeks of enrolment. Serum albumin ≥ 23 g/L within 2 weeks of enrolment.
10. Eastern Cooperative Oncology Group (ECOG) Performance Scale Score ≤ 2 measured within 2 weeks of enrolment.
11. Provide written informed consent prior to enrolment.

Group B (Maintenance Therapy) Inclusion Criteria:

1. Male or female ≥ 14 - 90 years of age.
2. Have previously received Lu-DOTA-TATE treatment under the SAP.
3. Life expectancy greater than 12 weeks from enrolment.
4. Serum creatinine ≤ 150 μmol/L, and a calculated (Cockcroft-Gault) or estimated glomerular filtration rate (GFR) of ≥ 50 mL/min measured within 2 weeks of enrolment.
5. Haemoglobin concentration ≥ 90 g/L; white blood cell (WBC) count ≥ 2 x 10^9/L; platelets ≥ 100 x 10^9/L measured within 2 weeks of enrolment.
6. Liver function tests (total bilirubin, alanine transaminase (ALT), aspartate transaminase (AST)) ≤ 3X the limit of normal measured within 2 weeks of enrolment. Serum albumin ≥ 23 g/L within 2 weeks of enrolment.
7. Eastern Cooperative Oncology Group (ECOG) Performance Scale Score ≤ 2 measured within 2 weeks of enrolment.
8. Provide written informed consent prior to enrolment.

Group A (Primary Therapy) Exclusion Criteria:

1. Have previously received Lu-DOTA-TATE therapy.
2. Potential for surgery with curative intent. Local surgery for symptomatic relief permitted as long as target lesion unaffected.
3. Major surgery within 12 weeks of enrolment. Minor surgeries such as removal of superficial skin lesions, laser eye surgery, cataract surgery, laparoscopic procedures and other procedures that are minimally invasive are permitted at the Investigator's discretion.
4. Liver embolization [transcatheter arterial embolization (TAE), TACE, or TARE] within 4 weeks of enrolment.
5. Radioisotope therapy within 12 weeks of enrolment.
6. Systemic therapy: mTOR inhibitors and tyrosine kinase inhibitors within 6 weeks of enrolment; chemotherapy and interferon within 8 weeks of enrolment.
7. Change in long-acting somatostatin analogues, dosage, or dosage frequency within 12 weeks of enrolment unless changes are required to manage uncontrolled symptoms.
8. Localized external beam irradiation with target lesion(s) in the radiation field. Other localized external beam therapy is permitted.
9. Known brain metastases unless these metastases have been treated and stabilized (confirmed by CT) for ≥ 4 months prior to enrolment
10. Uncontrolled diabetes mellitus defined as random glucose ≥ 2X the upper limit of normal (or HbA1c > 10%, if results available) within 12 weeks of enrolment.
11. Another significant medical, psychiatric or surgical condition uncontrolled by treatment, which may interfere with completion or conduct of the study (such as urinary incontinence, co-existing malignancies).
12. Pregnancy.
13. Breast feeding.
14. Prior radiation therapy to more than 25% of the bone marrow.
15. If, in the opinion of the investigator, other treatments are considered more appropriate than the investigational therapy, based on patient and disease characteristics.
16. Known allergy to somatostatin analogues or any components of the study medication.

Group B (Maintenance Therapy) Exclusion Criteria:

1. Another significant medical, psychiatric or surgical condition uncontrolled by treatment, which may interfere with completion or conduct of the study (such as urinary incontinence or co-existing malignancies).
2. Pregnancy.
3. Breast feeding.
4. Known allergy to somatostatin analogues or any components of the study medication.

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-04-29 (Actual); Primary Completion 2042-12 (Estimated); Study Completion 2042-12 (Estimated)

PRIMARY OUTCOMES:
Change in Tumour response of the target lesion(s) through end of treatment | At screening, 12-20 weeks after each treatment cycle, and 6 months and 1 year after the last treatment
  Tumor response of the target lesions(s) will be assessed by anatomic criteria in reference to RECIST 1.1 used in conjuction with lesion avidity on Nuclear Medicine scans, such as Lu-177 post-therapy scans, Octreoscan, [68]Ga-DOTATATE or [68]Ga-HA-DOTATATE PET, [18]F-FDG PET, [18]F-FDOPA PET, and/or others, as clinically indicated.
Median progression-free survival | Up to 1 year after last treatment
  Time from date of enrolment to the first documented target lesion progression or death due to any cause, which ever occurs first.
Lu-177 scan disease evaluation | Up to 3 days after each Lu-DOTA-TATE treatment
  A post-therapy Lu-177 scan will be conducted up to 3 days after each Lu-DOTA-TATE treatment to determine the intensity of tumour uptake of Lu-DOTA-TATE and the extent of tumour burden. Changes in Lu-177 scan data will also be used to stratify tumour response.
Change in tumour marker levels | At baseline, 12-20 weeks after each treatment cycle, and 6 months and 1 year after last treatment
  As clinically indicated, serum Chromogranin-A, urinary 5-HIAA, metanephrines, and/or other tumour markers will be collected at baseline, at each re-evaluation, at end of treatment, and at 6 months and 1 year after the last treatment. Tumour marker parameters will be recorded and all changes will be summarized.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 5 years after last treatment
  All participants will be evaluated for AE occurence from treatment 1 up to 5 years after the last treatment.
Change in haematology | At screening, within 2 weeks prior to at 6 weeks after each treatment, at each re-evaluation, and at 6 months and 1 year after last treatment.
  Blood samples will be analyzed for hemoglobin, platelet count, white blood cell count, lymphocyte count, and neutrophil count to monitor and record clinically significant out of range values that are indicative of toxicity. Samples will be collected at screening, within 2 weeks prior to each treatment, 6 weeks after each treatment, at each re-evaluation (12-20 weeks after treatments 4, 6, 8, and 10) and at 6 months and 1 year after the last treatment. Changes will be analyzed using descriptive statistics, and any identified adverse events will be tabulated and categorized according to CTCAE v.4.
Change in renal function | At screening, within 2 weeks prior to at 6 weeks after each treatment, at each re-evaluation, and at 6 months and 1 year after last treatment
  Blood samples will be analyzed for creatinine in order to calculate the glomerular filtration rate (GFR) and monitor and record clinically significant out of range values that are indicative of toxicity. Samples will be collected at screening, within 2 weeks prior to each treatment, 6 weeks after each treatment, at each re-evaluation (12-20 weeks after treatments 4, 6, 8, and 10) and at 6 months and 1 year after the last treatment. Changes will be analyzed using descriptive statistics, and any identified adverse events will be tabulated and categorized according to CTCAE v.4.
Change in liver function | At screening, within 2 weeks prior to at 6 weeks after each treatment, at each re-evaluation, and at 6 months and 1 year after last treatment
  Blood samples will be analyzed for total bilirubin, aspartate transaminase, and alanine transaminase to monitor and record clinically significant out of range values that are indicative of toxicity. Samples will be collected at screening, within 2 weeks prior to each treatment, 6 weeks after each treatment, at each re-evaluation (12-20 weeks after treatments 4, 6, 8, and 10) and at 6 months and 1 year after the last treatment. Changes will be analyzed using descriptive statistics, and any identified adverse events will be tabulated and categorized according to CTCAE v.4.
Median, 1, 2, 3, 4, and 5-year overall survival | Up to 5 years after last treatment
  Time from date of enrolment to date of death due to any cause or date of censoring at the last time the participant was known to be alive.
Change in Quality of Life (EORTC QLQ) | Prior to each treatment
  The European Organisation for Research Treatment of Cancer (EORTC) QLQ-C30 v.3 in conjunction with the supplementary module QLQ-GI.NET21 Quality of Life questionnaires will be administered prior to each treatment on the visit date. The core questionnaire and supplementary module will be scored according to the scoring manual, and changes analyzed to assess the effect of Lu-DOTA-TATE treatment on Quality of Life.
Change in Quality of Life (ESAS-r) | Prior to each treatment
  The Edmonton Symptom Assessment System Revised (ESAS-r) will be administered prior to each treatment on visit date. The questionnaire will be scored according to the scoring manual, and changes analyzed to assess the effect of Lu-DOTA-TATE treatment on Quality of Life.
Change in tumour biology (optional) | Up to 1 year after last treatment
  Subjects who have had surgery prior to or after Lu-DOTA-TATE therapy may have existing tumour tissue sample tested to characterize NET tumour biology and the effects of Lu-DOTA-TATE therapy on tumour cell function.

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Morrish, MD, PhD, Principal Investigator — Professor of Endocrinology and Oncology, University of Alberta, Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada